CLINICAL TRIAL: NCT03585465
Title: Metro-PD1: a Phase I/II Trial Evaluating Anti-PD1 (Nivolumab) in Combination With Metronomic Chemotherapy in Children and Teenagers With Refractory / Relapsing Solid Tumors
Brief Title: Nivolumab in Combination With Metronomic Chemotherapy in Paediatrics Refractory / Relapsing Solid Tumors
Acronym: Metro-PD1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Anticancer Fund, Belgium (Other); Bristol-Myers Squibb (Industry); CTD-CNO (Unknown); ECS-Progastrin SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metro-PD1-1708; 2024-513470-22-00 (EU CTIS Number)
Record Dates: First submitted 2018-06-14; First posted 2018-07-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Childhood Solid Tumor
MeSH Terms: interventions — Vinblastine; Cyclophosphamide; Capecitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A: Cyclophosphamide Vinblastine Nivolumab (Experimental): This arm was applicable to first stage, and is closed
  Interventions: Drug: Vinblastine; Drug: Cyclophosphamide; Drug: Nivolumab
- B: Capecitabine Nivolumab (Experimental): This arm was applicable to first stage, and is closed
  Interventions: Drug: Capecitabine; Drug: Nivolumab
- C: Cyclophosphamide Vinblastine Capecitabine (Experimental): This arm was applicable to first stage, and is closed
  Interventions: Drug: Vinblastine; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Nivolumab
- "Metronomic CT " (Experimental): metronomic chemotherapy selected at the end of first stage (C: Cyclophosphamide Vinblastine Capecitabine)
  This arm is applicable to second stage, and 43 patients are expected
  Interventions: Drug: Vinblastine; Drug: Cyclophosphamide; Drug: Capecitabine
- "Metronomic CT + Nivolumab" (Experimental): metronomic chemotherapy selected at the end of first stage (C: Cyclophosphamide Vinblastine Capecitabine) + Nivolumab
  This arm is applicable to second stage, and 43 patients are expected
  Interventions: Drug: Vinblastine; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Nivolumab

INTERVENTIONS:
Drug: Vinblastine — * Experimentals Arm A or C (First stage): 2 mg/m2/day IV, weekly per cycle, 28 days cycle
  * Experimental Arms Metronomic or Metronomic+Nivolumab (second stage): see C
  Arms: "Metronomic CT "; "Metronomic CT + Nivolumab"; A: Cyclophosphamide Vinblastine Nivolumab; C: Cyclophosphamide Vinblastine Capecitabine
Drug: Cyclophosphamide — * Arm A (First stage): 30 mg/m2/day PO, D1-4// D8-11// D15-18// D22-25 per cycle, 28 days cycle
  * Arm C (First stage): 30 mg/m2/day PO, D1-D4// D15-D18 per cycle, 28 days cycle
  * Metronomic or Metronomic+Nivolumab Arm (second stage): see C
  Arms: "Metronomic CT "; "Metronomic CT + Nivolumab"; A: Cyclophosphamide Vinblastine Nivolumab; C: Cyclophosphamide Vinblastine Capecitabine
Drug: Capecitabine — * Arm B (First stage): 400 to 600 mg/m2/day PO, all days per cycle, 28 days cycle
  * Arm C (First stage): 400 to 600 mg/m2/day PO, D8-D11// D22-D25 per cycle, 28 days cycle
  * Metronomic or Metronomic+Nivolumab Arm (second stage): see C
  Arms: "Metronomic CT "; "Metronomic CT + Nivolumab"; B: Capecitabine Nivolumab; C: Cyclophosphamide Vinblastine Capecitabine
Drug: Nivolumab — * Arm A, B or C (First stage): 3 mg/kg IV, D1 & D15 per cycle, 28 days cycle
  * Metronomic+Nivolumab Arm (second stage): 3 mg/kg IV, D1 & D15 per cycle, 28 days cycle
  Arms: "Metronomic CT + Nivolumab"; A: Cyclophosphamide Vinblastine Nivolumab; B: Capecitabine Nivolumab; C: Cyclophosphamide Vinblastine Capecitabine

SUMMARY:
The study is a two-stage trial:

1. First stage (closed - 16 patients recruited in France):

   Phase I feasibility trial to evaluate the safety of the combination of Nivolumab + metronomic chemotherapy considering three possible metronomic chemotherapy regimens
2. Second stage (opened - 86 patients expected in France and Belgium):

   Phase II randomized controlled balanced 1:1 open-label trial comparing the efficacy of the metronomic chemotherapy regimen selected at the end of the previous stage (arm C: cyclophosphamide, capecitabine, vinblastine), with or without nivolumab.
3. "Trans-MetroPD1" ancillary sub-study is partially implemented since April 2022, and proposed to patients participating to second stage

DETAILED DESCRIPTION:
1. First stage (closed):

   * Arm A: Nivolumab + Cyclophosphamide-Vinblastine
   * Arm B: Nivolumab + Capecitabin
   * Arm C: Nivolumab + Cyclophosphamide-Vinblastine + Capecitabin

   Arm A and Arm B have been allocated sequentially (A/B/A/B/A/B). Arm C has been opened, since arm A and Arm B were deemed safe.

   In each arm, the second patient was not recruited before the first patient has been observed for a 28-day duration.
2. Second stage (opened):

   Following the analysis of safety data from first stage, and according to IDMC's recommendations on December 2020, the metronomic chemotherapy selected for second stage was arm C: cyclophosphamide, capecitabine, vinblastine

   Randomization will be balanced 1:1, controlling for:
   * histological type: embryonal brain tumor, ependymoma, low-grade glioma, rhabdomyosarcoma, neuroblastoma, Ewing sarcoma, and other solid tumors after approval from coordinators,
   * and treating center, using a dynamic allocation of treatment (minimization program) with a random factor set at 0.8.
3. Trans-MetroPD1 is divided into 3 axes:

   * to evaluate the health-related quality of life
   * to measure the kinectis of progastrin/hPG80, a biomarker over-expressed in a wide range of cancers
   * to determine the distribution of immune cells within blood tissue

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically proven diagnosis of solid malignant tumor. Confirmed progressive or refractory disease despite standard therapy or for which no effective standard therapy exists
* Histologically proven diagnosis of: embryonal brain tumor ; ependymoma ; low-grade glioma (LGG) ; high-grade glioma (HGG) except diffuse Intrinsic Pontine glioma (DIPG) Supratentorial Diffuse Midline Glioma K27M mutated are eligible ; rhabdomyosarcoma ; neuroblastoma ; Ewing sarcoma ; and other solid tumors and after approval from coordinators (except DIPG, osteosarcoma, lymphoma), and confirmed progressive or refractory disease despite standard therapy or for which no effective standard therapy exists (this criterion is applicable to stage 2 only)
* Male and female subjects < 18 years of age at inclusion; patients of 18 years and older may be included after discussion with the sponsor if they had a pediatric recurrent/refractory malignancy diagnosed before the age of 18.
* Evaluable or measurable disease as defined by adequate standard imaging criteria for each patient's tumor type (see corresponding appendices for definition of evaluable and/or measurable lesions):

  * RANO criteria for patients with high grade glioma (HGG), who are eligible at stage 1 only
  * RAPNO criteria for patients with low grade glioma
  * WHO for other cerebral tumors
  * INRC criteria for patients with neuroblastoma (NB),
  * RECIST v1.1 for tumors other than cerebral tumors and neuroblastoma
* Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 70%. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy ≥ 3 months
* Adequate organ function:
* Hematologic criteria

  * Peripheral absolute neutrophil count (ANC) ≥ 1500/mm3 (unsupported)
  * White blood cells count ≥ 2500/mm3
  * Platelet count ≥ 100,000/mm3 (unsupported)
  * Hemoglobin ≥ 8.0 g/dL (transfusion is allowed)
* Cardiac function

  * Shortening fraction (SF) >29% (>35% for children < 3 years) and left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography (mandatory only for patients who have received cardiotoxic therapy).
  * Absence of QTc prolongation (QTc > 450 msec on baseline ECG, using the Fridericia correction [QTcF formula]) or other clinically significant ventricular or atrial arrhythmia.
* Renal and hepatic function

  * Serum creatinine < 1.5 x upper limit of normal (ULN) for age
  * Total bilirubin < 1.5 x ULN,
  * Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) < 3 x ULN;
  * aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT < 3 x ULN
* Able to comply with scheduled follow-up and with management of toxicity.
* Females of child bearing potential must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment.
* Sexually active patients must agree to use adequate and appropriate contraception while on study drug and for 6 months after stopping the study drug for young men, and for 12 months after stopping the study drug for young women
* Patients on stable doses of corticosteroids (≤0.25 mg/kg prednisolone or equivalent) for at least 7 days prior to receiving study drug may be included.
* Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.
* Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.
* Patients can have received prior treatment with antiPD1 or antiPDL1 if at least SD for 6 months or PR or CR was obtained.
* Patients with a known partial deficiency of dihydro-pyrimidine-deshydrogenase (DPD) activity are eligible, and must have an uracilemia value ≥16ng/ml and <150ng/ml
* Adult patient (or parents/legal representatives if patient is minor) understand the preparation process of soluble capecitabine, and are able to reconstitute oral solution of capecitabine at home

EXCLUSION CRITERIA:

* Leukemia
* Diagnosis of lymphoma, diffuse intrinsic pontine glioma or osteosarcoma (for stage 2 only)
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of corticosteroids or local CNS-directed therapy to control their CNS disease.
* Patients requiring high doses of corticosteroids >0.25mg/kg prednisolone or equivalent) or increasing doses of corticosteroids during the 7 days prior to receiving study drug.
* For patients with CNS tumor:

  o Evidence of > Grade 1 recent CNS hemorrhage on the baseline MRI scan.

  o Participants with bulky tumor on imaging are ineligible; bulky tumor is defined as: i) Tumor with any evidence of uncal herniation or severe midline shift ii) Tumor with diameter of > 6 cm in one dimension on contrast-enhanced MRI iii) Tumor that in the opinion of the investigator, shows significant mass effect
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
* Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening)
* Active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
* Active autoimmune disease requiring immunosuppressive treatment
* Known congenital immunodeficiency
* Presence of any NCI-CTCAE v5 grade ≥ 2 treatment-related extra-hematological toxicity with the exception of alopecia, ototoxicity or peripheral neuropathy.
* Systemic anticancer therapy within 21 days of the first study dose or 5 times its half-life, whichever is less, 6 weeks in case of nitrosourea.
* No clinical benefit with previous antiPD1 or antiPDL1 treatment (SD during a period inferior to 6 months, or PD).
* Previous myeloablative therapy with autologous hematopoietic stem cell rescue within 8 weeks of the first study drug dose.
* Allogeneic stem cell transplant within 3 months prior to the first study drug dose. Patients receiving any agent to treat or prevent graft-versus host disease (GVHD) post bone marrow transplant are not eligible for this trial.
* Radiotherapy (non-palliative) within 21 days prior to the first dose of drug (or within 6 weeks for therapeutic doses of MIBG or craniospinal irradiation).
* Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48 hour interval must be maintained before the first dose of the investigational drug is administered.
* Currently taking medications with a known risk of prolonging the QT interval or inducing Torsades de Pointes.
* Known hypersensitivity to any study drug or component of the formulation.
* Absence of effective contraception in patients of childbearing age
* Pregnant or nursing (lactating) females.
* Vaccination with live, attenuated vaccines within 4 weeks of the first dose of the study drugs except inactivated vaccines.
* Patient with a known complete absence of DPD activity; it is known that patients carrying some homozygous or heterozygous mutations of DPYD responsible for the complete or almost complete absence of enzymatic activity of DPD, are exposed to a maximum risk of life-threatening or fatal toxicity ; patients with a complete deficiency of DPD activity (uracilemia ≥150ng/ml) should not be included in the trial neither treated with capecitabine
* Patients with galactose intolerance, Lapp lactase deficiency or glucose or galactose malabsorption syndrome (rare hereditary diseases)
* Acute urinary tract infection, pre-existing hemorrhagic cystitis; obstruction of the urinary tract
* History of organ transplant
* Severe infections requiring parenteral antibiotic therapy
* Active tuberculosis
* History of interstitial lung disease

INCLUSION CRITERIA FOR TRANS-METROPD1

* Patient or parents/legal representative has/have given written informed consent to participate to all or part of Trans-MetroPD1 study
* If patient or parents/legal representative agrees to participate to the dosage of circulating progastrin only, patient body weight must be ≥ 8 kg to allow sample collection while respecting blood volume limits in paediatric population
* If patient or parents/legal representative agrees to participate to immune cells count only, or both immune cells count and dosage of circulating progastrin, patient body weight must be ≥ 54 kg to allow sample collection while respecting blood volume limits in paediatric population

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities according to the NCI-CTCAE V5 | Over the first chemotherapy cycle (28 days)
  First Stage Primary Outcome 3 metronomic CT are : A:Cyclophosphamide + Vinblastine B:Capecitabin C:Cyclophosphamide + Vinblastine + Capecitabin
Progression-free survival according appropriate criteria (RANO, RAPNO, WHO, INRC, RECIST v1.1). | up to 2 years
  Second Stage Primary Outcome Metronomic chemotherapy is the same as regimen selected at the end of the first stage

SECONDARY OUTCOMES:
Adverse events according to the NCI-CTCAE V5. | up to 2 years
  First Stage Secondary Outcome 1 & Second Stage Secondary Outcome 1
Tumor response in terms of complete/partial response or stable/progressive disease (using RANO, RAPNO, WHO, INRC, or RECIST v1.1) and overall survival | up to 2 years
  Second Stage Secondary Outcome 2
Dose-intensity for each drug (ratio between the computed dose-intensity, and the protocol dose-intensity) | up to 2 years
  First Stage Secondary Outcome 2 & Second Stage Secondary Outcome 3
Description of molecular profile (number of genetic alterations) on individual tumor ; the data will be collected from large-scale analysis programs performed in Europe (Mappyacts, France Genomic 2025) in agreement with the Sponsors | At study entrance
  Second Stage Secondary Outcome 4
Health Related Quality of Life using the age-appropriate KINDL-R questionnaire (self- and proxy-assessment) | from date of randomization until the date of first documented progression or date corresponding to the end of treatment, assessed up to 24 months
  Second Stage Ancillary Outcome 1
Dosage of circulating progastrine (hPG80) on blood-derived samples. | from date of randomization until the date of first documented progression or date corresponding to the end of treatment, up to 24 months
  Second Stage Ancillary Outcome 2
Counting of immune cells (number of: B cells, T cells, NK cells, dendritic cells subsets, and monocytes populations at each timepoint) on blood and blood-derived samples with flow cytometry analysis | At day-0, Day-8, Day-15, Day-28, Day-42, and until the date of first documented progression (assessed up to 24 months)
  Second Stage Ancillary Outcome 3

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBLOND, MD, Study Director — Centre Oscar Lambret; Nicolas ANDRE, MD, Study Director — CHU La Timone; Leen WILLEMS, MD, Study Director — University Hospital, Ghent
Locations (11):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc (CUSL), Brussels
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven
- France (8):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard (IHOPe), Lyon
  - Hôpital La Timone, AP-HM, Marseille
  - Hôpital d'Enfants - CHRU Nancy, Nancy
  - Hôpital Mère-Enfant, CHU Nantes, Nantes
  - Institut Curie, Paris
  - Hôpital de Hautepierre, CHRU Strasbourg, Strasbourg
  - Hôpital des Enfants - CHU Toulouse, Toulouse